CLINICAL TRIAL: NCT04272008
Title: A Study to Evaluate the Effects of Annovera™ and Tampon Co-Usage on the Pharmacokinetics of Segesterone Acetate and Ethinyl Estradiol
Brief Title: The Effects of Annovera™ and Tampon Co-Usage on the Pharmacokinetics of Segesterone Acetate and Ethinyl Estradiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TherapeuticsMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANNOV3454-3 PMR
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Contraception
Keywords: tampon; vaginal ring
MeSH Terms: interventions — segesterone acetate and ethinyl estradiol vaginal system

STUDY DESIGN:
Intervention Model Description: This is an open label, randomized, crossover PK study. Participants will be randomized to one of two treatment sequences. Each treatment sequence consists of two cycles of treatment - one with tampon use and one without tampon use. Tampon use will occur on Days 2 to 5 of contraceptive vaginal system (CVS) use and a new CVS will be used for each treatment cycle. Before starting Annovera use, each subject will use a combined oral contraceptive (COC) for one cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Annovera (alone) (Active Comparator): Annovera without tampon use
  Interventions: Drug: Segesterone Acetate and Ethinyl Estradiol
- Annovera with tampon use (Active Comparator): Annovera with tampon use
  Interventions: Drug: Segesterone Acetate and Ethinyl Estradiol; Other: Tampon

INTERVENTIONS:
Drug: Segesterone Acetate and Ethinyl Estradiol — Annovera taken alone
  Other Names: Annovera
Other: Tampon — Annovera with tampon use
  Arms: Annovera with tampon use

SUMMARY:
This study will evaluate the effect of Annovera and tampon co-usage on the pharmacokinetics (PK) of segesterone acetate (SA) and ethinyl estradiol (EE).

DETAILED DESCRIPTION:
This is an open label, randomized, crossover PK study. Participants will be randomized to one of two treatment sequences. Each treatment sequence consists of two cycles of treatment - one with tampon use and one without tampon use. Tampon use will occur on Days 2 to 5 of contraceptive vaginal system (CVS) use and a new CVS will be used for each treatment cycle. Before starting Annovera use, each subject will use a combined oral contraceptive (COC) for one cycle.

ELIGIBILITY:
Inclusion Criteria

All of the following criteria must be met for the participants to be eligible for the study:

1. Healthy women, sterile or at risk of becoming pregnant, inclusive of ages 18 to 35* years at the enrollment visit.
2. Intact uterus and both ovaries.
3. Prior history of regular menstrual cycles that usually occur every 28 ± 7 days when not using hormonal contraception; if postpartum or post-abortal, history of regular menstrual cycles of 21 to 35 days in length and resumption of at least one cycle with a cycle length consistent with her past cycles.
4. In the opinion of the Investigator, able to comply with the protocol, eg, live within the study site catchment area or within a reasonable distance from the study site.
5. Willing to use oral contraception for one month prior to the initial insertion of Annovera.
6. Willing to abstain from tampon use except during the prescribed time of the trial.
7. Willing to abstain from sexual intercourse during tampon use.
8. Signed informed consent prior to entry into the trial.

   * Upper age limit based on normal ovarian changes (ovarian reserve) prevalent in women with advancing age (> 35 years of age) that may alter patterns of follicle development and/or confound interpretations of data regarding patterns of follicle development

Exclusion Criteria

Contraindications for enrollment will be the same as those for use of CHCs and additional criteria important to the objectives of this study and include:

1. Known hypersensitivity to estrogens or progestins.
2. Pregnant, trying to become pregnant, or breastfeeding.
3. Known hypersensitivity to silicone rubber.
4. Undiagnosed abnormal vaginal bleeding.
5. Undiagnosed vaginal discharge, vaginal lesions or abnormalities. Participants diagnosed at screening with a chlamydia or gonococcus infection may be included in the trial following treatment; partner treatment is also recommended. Investigators should make a determination if participants are at high risk for reinfection, eg, multiple sex partners, untreated partner, and whether such participants can be included.
6. History of pelvic inflammatory disease since the participant's last pregnancy.
7. History of toxic shock syndrome.
8. In accordance with the Bethesda system of classification: Women with a current (within the last 20 months) abnormal Papanicolaou smear (Pap smear) suggestive of high-grade pre-cancerous lesion (s), including high grade squamous intraepithelial lesion.
9. Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring.
10. Women planning to undergo major surgery during the trial.
11. Women who smoke 15 cigarettes or more per day must be evaluated by the Principal Investigator (PI) for inclusion based on risk factors that would increase their risk for cardiovascular disease and thromboembolism, eg, lipid levels, glucose level, blood pressure (BP), body mass index (BMI), family history of cardiovascular disease at a young age.
12. Current or past thrombophlebitis or thromboembolic disorders.
13. History of venous thrombosis or embolism in a first-degree relative, < 55 years of age suggesting a familial defect in the blood coagulation system, which in the opinion of the PI, suggests that use of a hormonal contraceptive could pose a significant risk.
14. Cerebrovascular or cardiovascular disease.
15. History of retinal vascular lesions, unexplained partial or complete loss of vision.
16. Known or suspected carcinoma of the breast.
17. Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
18. Past history of any other carcinoma unless in remission for more than five years.
19. Current or history of medically diagnosed severe depression, which, in the opinion of the Investigator, could be exacerbated by the use of a hormonal contraceptive.
20. Has a Type D personality type as assessed by the DS14 test (Standard Assessment of Negative Affectivity, Social Inhibition and Type D Personality).
21. Headaches with focal neurological symptoms.
22. Severe constipation in the opinion of the Investigator.
23. History of cholestatic jaundice of pregnancy or jaundice with prior steroid use.
24. Benign or malignant liver tumors; active liver disease.
25. Diastolic BP > 85 mm Hg and/or systolic BP > 135 mm Hg after 5 to 10 minutes rest (at Screening).
26. Known or suspected alcoholism or drug abuse within their lifetime. aa. Elevated serum fasting clinical chemistry values or complete blood count (CBC) values designated clinically significant by the Investigator and/or medically qualified Sub-Investigator.

bb. Screening hemoglobin levels less than 12.5 g/dL or hematocrit less than 38%.

cc. Participation in another clinical trial involving an investigational drug within the last 30 days (prior to Screening). dd. BMI > 29 kg/m2. ee. Use of liver enzyme inducers on a regular basis. ff. Use of monthly injectable contraceptives, unless suspended 2 months before initiation of the treatment. Use of Depo-Provera® [depot medroxyprogesterone acetate] unless suspended 9 months before treatment.

gg. Current use of implanted hormonal contraceptives, including Mirena® [progestin containing intrauterine system], Jadelle®, Norplant®, Implanon® or Nexplanon (if now available in the USA).** hh. Known HIV, Hepatitis B or Hepatitis C infection. ii. History of frequent vaginal infections in the opinion of the PI. jj. Use of any oral medications or supplements during the trial that could interfere with the metabolism of the contraceptive hormones. Use of any vaginal preparations during Treatment Cycle 1 or Treatment Cycle 2. Use of any medication during the study must be reviewed and approved by the Medical Monitor

*Women using non-hormonal intrauterine devices are permitted to enroll in the study.

**Participants using any of the implanted hormonal methods who request removal for reasons unrelated to the purpose of enrollment in this study may be considered for participation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
The effect of Annovera and tampon co-use on area-under-the-curve (AUC) of Segesterone acetate and ethinyl estradiol (Days 2 to 3) | Days 2 to 3
  AUC for 24 hours

SECONDARY OUTCOMES:
The effect of Annovera and tampon co-use on area-under-the-curve (AUC) of Segesterone acetate and ethinyl estradiol (Days 2 to 5) | Days 2 to 5
  AUC for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mirkin, MD, Study Chair — TherapeuticsMD
Locations (2):
- University of Pennsylvania Women's Health Clinical Research Center, Philadelphia, Pennsylvania, United States
- Syneos Health, Québec, Quebec, Canada